CLINICAL TRIAL: NCT03695614
Title: Cognitive Remediation Therapy for Participants With Late-Life Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Angela Golas, Geriatric Psychiatrist, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 083/2017
Record Dates: First submitted 2018-09-03; First posted 2018-10-04 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia; Cognitive Remediation; Late Life Schizophrenia; Functional Impairment; Cognitive Deficit
MeSH Terms: conditions — Schizophrenia; Cognition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Remediation (Experimental): CR is a form of group therapy that uses a hybrid approach of restorative and strategy based methods to improve areas of cognition (ie. attention, memory, processing speed and learning) through the use of computerized exercises. CR is administered in groups consisting of 2-8 participants and one or two therapists. The CR groups meet twice per week for two hours per session over twelve weeks, for a total of 24 sessions.
  Interventions: Other: Cognitive Remediation Therapy

INTERVENTIONS:
Other: Cognitive Remediation Therapy — Cognitive Remediation is a well-established psychotherapy that aims to improve neurocognitive abilities such as memory performance, executive functioning, processing speed, and attention.

SUMMARY:
Cognitive Remediation (CR) involving restorative and strategy-based methods has been previously validated in a pilot study for late life schizophrenia (LLS), where CR demonstrated a moderate effect on overall cognition. This study proposes to study the efficacy of CR in a larger cohort of participants with LLS and to assess the interaction of medication management with CR on cognitive outcomes. Eligible participants will receive CR during 12 weeks. CR consists of a series of computerized exercises targeting various cognitive functions, such as memory, attention and processing speed. It will be administered during facilitated group sessions consisting of 4-6 people.

The study will recruit 40 participants with the aim to enroll 30 LLS participants age 55 or older who will undergo the CR intervention for two, 2-hour weekly classes over 12 weeks (24 classes in total). There will be baseline assessments (clinical and NP) prior to enrollment in the classes. In order to assess whether there has been a change in cognition, and some of the assessments will be repeated after the 12-week intervention.

DETAILED DESCRIPTION:
Thirty late life schizophrenia (LLS) participants, age 55 and over, will undergo the CR intervention after completion of the baseline assessments. CR is a group-based psychotherapy that will consist of two, 2-hour weekly therapist-guided classes over 12 weeks, with a half-hour lunch break. The 24 classes are divided into two iterations of 12 exercises each, repeated twice. CR consists of four techniques: (1) didactic teaching on the relevance of cognition for everyday functioning and the association between cognitive strategies and enhanced functioning (2) computerized drills targeting different cognitive domains, (3) in-class strategic monitoring to enhance metacognitive skills, and (4) discussion of the generalization of cognitive skills to daily life. The Brain Gym includes electronic tablets for participant use both during classroom sessions in addition to elective, drop-in practice sessions offered three times per week. Each group will consist of 4-6 participants. A group will be started once four to six consecutively referred participants complete baseline assessments. Each class is self-contained and the first class is always introductory to CR in order to enhance the comfort level with the computer equipment and program.

Each of the 24 classes will have one, 5-10 minute block of didactic teaching, two 45-minute blocks of drill-and-practice of the online exercises, and a 20-minute lunch break. Exercises are delivered via Scientific Brain Training (SBT) Pro (2009). Computer exercises are designed to be enjoyable and reinforcing, with the difficulty level gradually increasing over time. The therapists optimize competency and motivation by individualizing the exercises for each participant. The difficulty level parameters are manually titrated according to exercise adherence and difficulty level progression, targeting 80 percent accuracy in order to optimize competency and motivation. In order to optimize learning and retention outside of weekly classes, participants are encouraged to return to the computer lab for ongoing practice of the online exercises, targeting 40 minutes of homework exercises per weekday for a total target of 200 minutes per week. Online logs allow for monitoring the time spent completing the computer exercises. The therapists review the online logs on a weekly basis with the participants at the end of the didactic class and before planning the homework for the following week. Participants' successful completion of a given exercise to the highest difficulty level is charted in the Brain Gym using their anonymized computer log-in name to serve as positive reinforcement and recognition of their achievement while maintaining privacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55 years and above. The rationale of age cutoff of 55 is that this age is considered a typical geriatric age cutoff for participants with LLS.
2. Any race or ethnicity.
3. Females and males.
4. Meets DSM-V criteria for a current diagnosis of schizophrenia or schizoaffective disorder.
5. Clinically stable as operationalized by (1) having not been admitted to a psychiatric hospital within the 3 months prior to assessment, (2) having had no change in antipsychotic medication dosage within the 4 weeks prior to assessment, and (3) and ascertained to be clinically and medically stable by one of the study psychiatrists.
6. Willingness and ability to speak English
7. Willingness to provide informed consent
8. Corrected visual ability that enables reading of newspaper headlines and corrected hearing capacity that is adequate to respond to a raised conversational voice.

Exclusion Criteria:

1. Meets criteria for a cognitive disorder secondary to a neurological or other medical disorder
2. Diagnosis of bipolar disorder or current major depressive episode
3. Meets diagnostic criteria for substance use or dependence within the 6 months prior to the initial assessment except for caffeine or nicotine
4. Electroconvulsive Therapy (ECT) within 6 months of initial assessment

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Assess the effect of CR on cognitive performance as indicated by total Montreal Cognitive Assessment (MoCA) scores | approximately 12 weeks after the baseline
  Total score out of 30 possible points, with 30/30 indicating best possible score

SECONDARY OUTCOMES:
Assess effect of Cognitive Remediation (CR) on tolerability of CR according to the percentage of participants completing the 12-week course | approximately 12 weeks after the baseline
  Range of 0-100% individuals completing, with 100% completers indicating best possible outcome.
Change in general, positive, and negative symptoms of Schizophrenia as assessed by the Positive and Negative Syndrome Scale | At baseline and approximately 12 weeks after the baseline
  Total score range of 30-210, 30 indicating the best possible score
Change in depressive symptoms as assessed by the Calgary Depression Scale for Schizophrenia | At baseline and approximately 12 weeks after the baseline
  Score range of 0-27, 0 indicating the best possible score
Change in visuospatial/executive domains of cognition as assessed by the Trail making Test B and A | At baseline and approximately 12 weeks after the baseline
  Scored via number of correct moves ranging from 0-24, 24 indicating best possible score. Also scored via number of errors made, ranging from 0-24, 0 indicating best possible score
Change in immediate memory, visuospatial/constructional cognition, language, attention, and delayed memory as assessed by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | At baseline and approximately 12 weeks after the baseline
  Subscales include List Learning (0-40, 40 indicating best possible score) and Story Memory (0-24, 24 indicating best possible score) for testing of immediate memory. Figure Copy (0-20, 20 indicating best possible score) and Line Orientation (0-20, 20 indicating best possible score) for testing of visuospatial/constructional cognition. Picture Naming (0-10, 10 indicating best possible score) and Semantic Fluency (4-40, 40 indicating best possible score) for testing of language. Digit Span (0-16, 16 indicating best possible score) and Coding (0-89, 89 indicating best possible score) for testing of attention. List Recall (0-10, 10 indicating best possible score), List Recognition (0-20, 20 indicating best possible score), Story Recall (0-12, 12 indicating best possible score), and Figure Recall (0-20, 20 indicating best possible score) for testing of delayed memory.
Change in executive functioning and planning ability as assessed by the Tower of London | At baseline and approximately 12 weeks after the baseline
  Change in executive functioning and planning ability as assessed by the Tower of London
Change in verbal working memory as assessed by the Letter Number Span | At baseline and approximately 12 weeks after the baseline
  Score range of 0-24, 24 indicating best possible score
Change in visual working memory as assessed by the Wechsler Memory Scale Spatial Span | At baseline and approximately 12 weeks after the baseline
  Scored via number of correct forward items (0-16, 16 indicating best possible score). Also scored via number of correct backwards items (0-16, 16 indicating best possible score)
Degree of anticholinergic burden of medication used by our participants, quantified by the Anticholinergic Burden Scale (ACB) | At baseline
  A total ACB scale score of three or more is considered clinically relevant

CONTACTS AND LOCATIONS:
Overall Officials: Angela Golas, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada